CLINICAL TRIAL: NCT00457821
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study of VX-770 to Evaluate Safety, Pharmacokinetics, and Biomarkers of CFTR Activity in Cystic Fibrosis (CF) Subjects With Genotype G551D
Brief Title: Safety Study of Ivacaftor in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX06-770-101
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis
Keywords: G551D mutation; Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ivacaftor Group A (Experimental): Subjects in Part 1 who first received 25 mg or 75 mg of ivacaftor every 12 hours (q12h) for 14 days, then crossed over to receive the alternate dose for another 14 days.
  Interventions: Drug: Ivacaftor 25 mg/75 mg
- Ivacaftor Group B (Experimental): Subjects in Part 1 who first received 75 mg or 150 mg of ivacaftor q12h for 14 days then crossed over to receive the alternate dose for another 14 days.
  Interventions: Drug: Ivacaftor 75 mg/150 mg
- Ivacaftor Group C (Experimental): Subjects in Part 2 who received 150 mg or 250 mg of ivacaftor q12h for 28 days.
  Interventions: Drug: Ivacaftor 150 mg or 250 mg
- Placebo (Placebo Comparator): Subjects who received placebo in Part 1 and subjects who received placebo in Part 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor 25 mg/75 mg — 25 mg or 75 mg q12h for a total of 28 days (Part 1)
  Other Names: VX-770
  Arms: Ivacaftor Group A
Drug: Ivacaftor 75 mg/150 mg — 75 mg or 150 mg q12h for a total of 28 days (Part 1)
  Other Names: VX-770
  Arms: Ivacaftor Group B
Drug: Ivacaftor 150 mg or 250 mg — 150 mg or 250 mg of ivacaftor q12h for 28 days (Part 2)
  Other Names: VX-770
  Arms: Ivacaftor Group C
Drug: Placebo — Given q12h for 28 days each in Part 1 and Part 2 of the study
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of ivacaftor in patients with cystic fibrosis (CF) who were aged 18 years or older and have a G551D mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. Ivacaftor is a potent and selective CFTR potentiator of wild-type, G551D, F508del, and R117H forms of human CFTR protein. Potentiators are pharmacological agents that increase the chloride ion transport properties of the channel in the presence of cyclic AMP-dependent protein kinase A (PKA) activation.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, cross-over, multiple dose study of up to 28 days of dosing, in subjects with cystic fibrosis (CF) who have a G551D-CTFR gene mutation. Enrollment of 39 subjects occurred at 15 centers in the US, Canada, and Germany.

The study was conducted in 2 parts:

* Part 1 consisted of Group A and Group B. Subjects in Group A (10 subjects) were randomized to receive 25 mg of ivacaftor every 12 hours [q12h] (4 subjects), 75 mg of ivacaftor q12h (4 subjects), or placebo (2 subjects) for 14 days. Following a 7- to 28-day washout period, subjects who received active study drug crossed over to the alternate dose strength of ivacaftor for an additional 14 days. Placebo subjects continued to receive placebo for an additional 14 days. Subjects in Group B (10 subjects) were randomized to receive 75 mg of ivacaftor q12h (4 subjects), 150 mg of ivacaftor q12h (4 subjects), or placebo (2 subjects) for 14 days. Following a 7- to 28-day washout period, the subjects who received active study drug crossed over to the alternate dose strength of ivacaftor for an additional 14 days. Placebo subjects continued to receive placebo for an additional 14 days.
* Part 2 consisted of Group C; these subjects did not participate in Part 1. Subjects were randomized to receive 150 mg of ivacaftor q12h (7 subjects), 250 mg of ivacaftor q12h (7 subjects), or placebo (4 subjects) for a total of 28 days. Ivacaftor doses studied in Part 2 were selected following an interim pharmacokinetic/pharmacodynamic (PK/PD) and statistical analyses of data from Part 1. The 2 doses selected for Part 2 were anticipated to enable better definition of the optimal therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Weighing at least 40 kg
* Confirmed diagnosis of cystic fibrosis (CF) and G551D mutation in at least 1 allele
* Forced expiratory volume in 1 second (FEV1) of at least 40% of predicted normal for age, gender, and height
* Willing to remain on stable medication regimen for the duration of study participation
* No significant clinical laboratory abnormalities, not pregnant, and willing to use at least 2 highly effective birth control methods during Part 1 and 1 highly effective birth control method during Part 2 of the study
* No clinically significant abnormalities that would have interfered with the study assessments, as judged by the investigator

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering study drug to the subject
* Ongoing acute respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 14 days of Day 1 of the study
* History of alcohol, medication or illicit drug abuse within one year prior to Day 1
* Abnormal liver function ≥ 3x the upper limit of normal
* History of abnormal renal function (creatinine clearance < 50 mL/min using Cockcroft-Gault equation)
* History of solid organ or hematological transplantation
* Pregnant or breast-feeding (for women)
* Ongoing participation in another therapeutic clinical trial, or prior participation in an investigational drug study without appropriate washout
* Concomitant use of any inhibitors or inducers of cytochrome P450 3A4 (CYP3A4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (15):
- United States (13):
  - University of Alabama Hospital, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - The Children's Hospital, Aurora, Colorado
  - Roy J. and Lucille A. Carver College of Medicine, The University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Pulmonary and Critical Care Medicine, Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital of Boston, Boston, Massachusetts
  - Division of Pulmonary, Allergy and Critical Care Medicine, University of Minnesota, Minneapolis, Minnesota
  - Cystic Fibrosis Pulmonary Research and Treatment Center, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pulmonary Critical Care, University of Washington, Seattle, Washington
- Division of Gastroenterology, Hepatology and Nutrition, The Hospital for Sick Children, Toronto, Ontario, Canada
- CF Clinic, Pediatric Pulmonology and Neonatology, Medical School of Hannover, Straße, Hannover, Germany

REFERENCES:
- [Result] Accurso FJ, Rowe SM, Clancy JP, Boyle MP, Dunitz JM, Durie PR, Sagel SD, Hornick DB, Konstan MW, Donaldson SH, Moss RB, Pilewski JM, Rubenstein RC, Uluer AZ, Aitken ML, Freedman SD, Rose LM, Mayer-Hamblett N, Dong Q, Zha J, Stone AJ, Olson ER, Ordonez CL, Campbell PW, Ashlock MA, Ramsey BW. Effect of VX-770 in persons with cystic fibrosis and the G551D-CFTR mutation. N Engl J Med. 2010 Nov 18;363(21):1991-2003. doi: 10.1056/NEJMoa0909825. PMID 21083385
- [Derived] Accurso FJ, Van Goor F, Zha J, Stone AJ, Dong Q, Ordonez CL, Rowe SM, Clancy JP, Konstan MW, Hoch HE, Heltshe SL, Ramsey BW, Campbell PW, Ashlock MA. Sweat chloride as a biomarker of CFTR activity: proof of concept and ivacaftor clinical trial data. J Cyst Fibros. 2014 Mar;13(2):139-47. doi: 10.1016/j.jcf.2013.09.007. PMID 24660233
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 started on 10 May 2007 (signing of first informed consent). After obtaining consent, Part 1 screening evaluations were completed during Day -28 to Day -2. Part 2 started on 28 May 2008 (signing of first informed consent). Part 2 screening evaluations were also completed during Day -28 to Day -2 before the first dose of study drug.
Pre-assignment Details: In Part 1, 21 subjects were randomized but 1 subject was excluded prior to dosing because the subject needed a protocol-prohibited medication. In Part 2, 20 subjects were randomized but 1 subject withdrew consent to the study prior to dosing.
Groups:
- Part 1: Placebo: Part 1: placebo every 12 hours (q12h); 14 days/14 days.
- Part 1: 25 mg/75 mg: Part 1: Ivacaftor (25 mg/75 mg) every 12 hours (q12h); 14 days/14 days.
- Part 1: 75 mg/25 mg: Part 1: Ivacaftor (75 mg/25 mg) every 12 hours (q12h); 14 days/14 days.
- Part 1: 75 mg/150 mg: Part 1: Ivacaftor (75 mg/150 mg) every 12 hours (q12h); 14 days/14 days.
- Part 1: 150 mg/75 mg: Part 1: Ivacaftor (150 mg/75 mg) every 12 hours (q12h); 14 days/14 days.
- Part 2: 150 mg: Part 2: Ivacaftor (150 mg) q12h; 28 days
- Part 2: 250 mg: Part 2: Ivacaftor (250 mg) q12h; 28 days
- Part 2: Placebo: Part 2: placebo q12h; 28 days
Period: Part 1
Arm/Group | Part 1: Placebo | Part 1: 25 mg/75 mg | Part 1: 75 mg/25 mg | Part 1: 75 mg/150 mg | Part 1: 150 mg/75 mg | Part 2: 150 mg | Part 2: 250 mg | Part 2: Placebo
Started | 4 (Number of subjects randomized) | 4 (Number of subjects randomized) | 5 (Number of subjects randomized) | 4 (Number of subjects randomized) | 4 (Number of subjects randomized) | 0 (Arm in Part 2 only) | 0 (Arm in Part 2 only) | 0 (Arm in Part 2 only)
Completed | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Placebo | Part 1: 25 mg/75 mg | Part 1: 75 mg/25 mg | Part 1: 75 mg/150 mg | Part 1: 150 mg/75 mg | Part 2: 150 mg | Part 2: 250 mg | Part 2: Placebo
Started | 0 (Arm in Part 1 only) | 0 (Arm in Part 1 only) | 0 (Arm in Part 1 only) | 0 (Arm in Part 1 only) | 0 (Arm in Part 1 only) | 8 (All subjects who received at least 1 dose of study drug (ivacaftor).) | 7 (All subjects who received at least 1 dose of study drug (ivacaftor).) | 5 (All subjects who received at least 1 dose of study drug (placebo).)
Completed Study Drug Treatment | 0 | 0 | 0 | 0 | 0 | 8 | 7 (1 subject missed a 250-mg dose of ivacaftor on Day 28 of Part 2.) | 4
Completed | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: 25 mg/75 mg | Part 1: 75 mg/25 mg | Part 1: 75 mg/150 mg | Part 1: 150 mg/75 mg | Part 2: 150 mg | Part 2: 250 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 4 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 34.5 (14.66) | 33.5 (12.50) | 38.5 (11.82) | 26.3 (7.85) | 23.5 (6.45) | 25.6 (7.98) | 26.0 (7.07) | 26.8 (10.69) | 28.7 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 3 | 3 | 5 | 3 | 1 | 20
  Male | 2 | 1 | 4 | 1 | 1 | 3 | 4 | 3 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 4 | 39
Weight [Mean (Standard Deviation); unit: kilograms] | 70.05 (16.507) | 66.05 (12.628) | 73.43 (14.366) | 57.48 (8.663) | 59.35 (18.401) | 61.19 (9.857) | 64.46 (13.027) | 63.50 (7.391) | 64.1 (12.42)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 24.195 (3.2002) | 22.455 (2.3133) | 23.653 (3.6216) | 20.960 (2.2522) | 20.788 (4.1527) | 21.896 (0.9770) | 22.703 (1.3980) | 22.035 (0.6999) | 22.3 (2.37)
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percentage of volume in liters] — Percent predicted for age, gender, and height.
  percentage of volume in liters | 64.902 (22.6821) | 71.073 (27.2307) | 54.885 (9.6772) | 68.284 (24.7014) | 49.270 (7.5615) | 70.443 (25.4442) | 72.674 (21.5223) | 79.351 (28.7018) | 67.3 (22.17)
Genotype [Number; unit: participants]
  G551D/1078 DEL T | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  G551D/DELTA F508 | 3 | 4 | 4 | 2 | 3 | 7 | 5 | 4 | 32
  G551D/G551D | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  G551D/N1303K | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  G551D/R553X | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  G551D/3849 AND 10KBC | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  G551D/6214 + 1G > 7T | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  G551D/G542X | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (Combined Part 1 and Part 2)
Description: Adverse event data were collected up to the follow-up visit (5 to 9 days after last dose of study drug). Serious adverse events that were ongoing at the follow-up visit were followed until the event resolved, returned to baseline, or was determined to be a stable or chronic condition.
Time Frame: Baseline to Follow-up
Population: All randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Number; unit: participants
Groups:
- Placebo: All subjects given placebo in Part 1 (n=4) and Part 2 (n=4)
- Ivacaftor: All subjects given Ivacaftor in Part 1 (n=16) and Part 2 (n=15)
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 8 | 31
participants
  Subjects with AEs | 7 | 26
  Subjects with Related or Possibly Related AEs | 3 | 13
  Subjects with SAEs | 0 | 1
  Subjects with Related or Possibly Related SAEs | 0 | 0

2. Secondary Outcome: Change From Baseline in Nasal Potential Difference (Combined Part 1 and Part 2)
Description: The transepithelial nasal potential difference (NPD) is a direct measure of transepithelial ion transport. NPD under conditions of zero chloride concentration perfusion solution in the presence of isoproterenol was of primary interest.
Time Frame: 14 days and 28 days
Population: Due to the crossover design in Part 1, subjects were counted once for each period; therefore, the 4 unique subjects who received placebo were counted as 8 subjects in the analyses for Part 1.
Measure: Least Squares Mean (95% Confidence Interval); unit: millivolts
Groups:
- Placebo: All subjects given placebo every 12 hours (q12h) in Part 1 (n=4) and Part 2 (n=4)
- 25 mg Ivacaftor q12h: All subjects given the 25 mg dose q12h in Group A in Part 1 (n=4 x 2).
- 75 mg Ivacaftor q12h: All subjects given the 75 mg dose q12h in Group A (n=4 x 2) and Group B (n=4 x 2) in Part 1.
- 150 mg Ivacaftor q12h: All subjects given the 150 mg dose q12h in Group B in Part 1 (n=4 x 2) and Group C in Part 2 (n=8).
- 250 mg Ivacaftor q12h: All subjects given the 250 mg dose q12h in Group C (n=7) in Part 2.
Arm/Group | Placebo | 25 mg Ivacaftor q12h | 75 mg Ivacaftor q12h | 150 mg Ivacaftor q12h | 250 mg Ivacaftor q12h
Number analyzed (Participants) | 12 | 7 | 15 | 16 | 7
millivolts
  Zero Chloride + Isoproterenol, Day 14 | -0.3 [-3.5 to 2.9] | -1.4 [-5.2 to 2.4] | -4.4 [-7.0 to -1.8] | -4.6 [-7.2 to -2.0] | -7.6 [-11.7 to -3.5]
  Zero Chloride + Isoproterenol, Day ≥ 14 | -0.5 [-4.1 to 3.1] | -1.3 [-5.2 to 2.6] | -4.5 [-7.3 to -1.7] | -5.3 [-7.9 to -2.6] | -8.4 [-12.3 to -4.5]
  Amiloride, Day 14 | 0.3 [-5.2 to 5.9] | -0.1 [-6.1 to 5.8] | -4.2 [-8.3 to 0.0] | -9.9 [-14.2 to -5.6] | -5.5 [-12.2 to 1.1]
  Amiloride, Day ≥ 14 | -0.7 [-5.5 to 4.1] | -0.3 [-6.8 to 6.2] | -3.7 [-8.4 to -1.0] | -8.8 [-12.8 to -4.8] | -4.0 [-9.2 to 1.2]
Statistical Analysis 1: Comparison: Placebo vs 25 mg Ivacaftor q12h vs 75 mg Ivacaftor q12h vs 150 mg Ivacaftor q12h vs 250 mg Ivacaftor q12h; Within-dose group and between-dose group analyses were performed, using a linear mixed effect model with baseline, dose, and period as fixed effects and subject as a random effect; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — There was no adjustment for multiple comparisons

3. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second [FEV1] (Combined Part 1 and Part 2)
Description: Spirometry is a standardized assessment to evaluate lung function that is the most widely used endpoint in cystic fibrosis studies.
  Relative change reflects the percent change from the baseline values [100% * (X-Y)/Y], where X and Y are post-baseline and baseline values, respectively.
Time Frame: 14 days and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted (%)
Arm/Group | Placebo | 25 mg Ivacaftor q12h | 75 mg Ivacaftor q12h | 150 mg Ivacaftor q12h | 250 mg Ivacaftor q12h
Number analyzed (Participants) | 10 | 7 | 15 | 16 | 7
percent predicted (%)
  Absolute Change from Baseline, Day 14 | 0.5 [-3.4 to 4.5] | 2.7 [-1.8 to 7.1] | 5.1 [2.0 to 8.3] | 6.9 [3.9 to 10.0] | 8.4 [3.7 to 13.2]
  Absolute Change from Baseline, Day ≥ 14 | 2.1 [-1.3 to 5.6] | 2.5 [-1.3 to 6.2] | 5.3 [2.4 to 8.1] | 6.9 [4.4 to 9.5] | 6.7 [3.1 to 10.3]
  Relative Change from Baseline, Day 14 | 2.0 [-4.8 to 8.9] | 4.7 [-2.7 to 12.2] | 9.5 [4.1 to 14.8] | 10.8 [5.6 to 15.9] | 12.0 [3.8 to 20.1]
  Relative Change from Baseline, Day ≥ 14 | 3.3 [-2.4 to 9.1] | 4.1 [-1.9 to 10.1] | 9.3 [4.7 to 13.9] | 10.6 [6.5 to 14.8] | 9.4 [3.4 to 15.4]
Statistical Analysis 1: Comparison: Placebo vs 25 mg Ivacaftor q12h vs 75 mg Ivacaftor q12h vs 150 mg Ivacaftor q12h vs 250 mg Ivacaftor q12h; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — There was no adjustment for multiple comparisons

4. Secondary Outcome: Change From Baseline in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) Score (Part 2 Only)(Respiratory Domain Score)
Description: The CFQ-R is a health-related quality of life measure for subjects with cystic fibrosis. Each domain is scored from 0 (worst) to 100 (best). A difference of at least 4 points in the respiratory domain score of the CFQ-R is considered a minimal clinically important difference (MCID).
Time Frame: 14 days and 28 days
Population: Part 2 is a parallel study. Subjects were counted only once for each treatment group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects given placebo every 12 hours (q12h) for 28 days.
- 150 mg Ivacaftor q12h: Subjects given 150 mg of ivacaftor q12h for 28 days.
- 250 mg Ivacaftor q12h: Subjects given 250 mg of ivacaftor q12h for 28 days.
Arm/Group | Placebo | 150 mg Ivacaftor q12h | 250 mg Ivacaftor q12h
Number analyzed (Participants) | 4 | 8 | 7
score on a scale
  Baseline Respiratory Domain Score | 70.8 (21.5) | 68.8 (23.9) | 73.0 (8.7)
  Change from Baseline in Respiratory Score, Day 14 | 2.8 (7.2) | 6.3 (6.9) | 5.6 (7.9)
  Change from Baseline in Respiratory Score, Day 28 | 2.8 (7.2) | 6.9 (6.5) | 11.9 (14.1)

5. Secondary Outcome: Change From Baseline in Maximum Sweat Chloride Concentration (Combined Part 1 and Part 2)
Description: The sweat chloride (quantitative pilocarpine iontophoresis) test is a standard diagnostic tool for cystic fibrosis (CF), serving as an indicator of cystic fibrosis transmembrane conductance regulator (CFTR) activity.
Time Frame: 14 days and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter
Arm/Group | Placebo | 25 mg Ivacaftor q12h | 75 mg Ivacaftor q12h | 150 mg Ivacaftor q12h | 250 mg Ivacaftor q12h
Number analyzed (Participants) | 12 | 8 | 14 | 16 | 7
millimoles per liter
  Change from Baseline in Sweat Chloride, Day 14 | 2.0 [-9.1 to 13.1] | -33.8 [-43.4 to -24.2] | -42.0 [-49.9 to -34.1] | -46.0 [-53.9 to -38.2] | -27.1 [-39.7 to -14.6]
  Change from Baseline in Sweat Chloride, Day ≥14 | 4.9 [-5.3 to 15.0] | -32.9 [-41.7 to -24.2] | -40.8 [-48.1 to -33.5] | -44.2 [-51.1 to -37.3] | -28.2 [-39.0 to -17.4]
Statistical Analysis 1: Comparison: Placebo vs 25 mg Ivacaftor q12h vs 75 mg Ivacaftor q12h vs 150 mg Ivacaftor q12h vs 250 mg Ivacaftor q12h; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — There was no adjustment for multiple comparisons

6. Primary Outcome: Number of Adverse Events (Combined Part 1 and Part 2)
Description: as for outcome 1
Time Frame: Baseline to Follow-up
Population: All randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Number; unit: events
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 8 | 31
events
  Number of Adverse Events (AEs) | 32 | 179
  Number of Related or Possibly Related AEs | 11 | 40
  Number of Serious Adverse Events (SAEs) | 0 | 2
  Number of Related or Possibly Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to the follow-up visit (5 to 9 days after last dose of study drug).
Arm/Group | Placebo | 25 mg Ivacaftor q12h | 75 mg Ivacaftor q12h | 150 mg Ivacaftor q12h | 250 mg Ivacaftor q12h
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 1/16 | 0/7
Other Adverse Events (participants affected / at risk) | 7/8 | 4/8 | 13/16 | 13/16 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 25 mg Ivacaftor q12h (N=8) | 75 mg Ivacaftor q12h (N=16) | 150 mg Ivacaftor q12h (N=16) | 250 mg Ivacaftor q12h (N=7)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — CF exacerbations were coded as "cystic fibrosis lung."
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 25 mg Ivacaftor q12h (N=8) | 75 mg Ivacaftor q12h (N=16) | 150 mg Ivacaftor q12h (N=16) | 250 mg Ivacaftor q12h (N=7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (3) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sputum decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Painful defaecation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (4) | 0 (0)
Catheter related complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) — CF exacerbations were coded as "cystic fibrosis lung."
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital pruritus female (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days